CLINICAL TRIAL: NCT03838614
Title: Rhythmical Auditory Stimulation Gait Training and Muscle Power Training for Primary School Children With Developmental Coordination Disorder: A Randomized Controlled Trial
Brief Title: Gait and Muscle Power Training for Children With Developmental Coordination Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Developmental Coordination Disorder
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RAS-MPT group (Experimental): Rhythmical auditory stimulation gait training and muscle power training group
  Interventions: Behavioral: Rhythmical auditory stimulation gait training and muscle power training (RAS-MPT)
- RAS group (Experimental): Rhythmical auditory stimulation gait training group
  Interventions: Behavioral: Rhythmical auditory stimulation gait training (RAS)
- MPT group (Experimental): Muscle power training group
  Interventions: Behavioral: Muscle power training (MPT)
- Control group (Other): Usual care group
  Interventions: Other: Controls

INTERVENTIONS:
Behavioral: Rhythmical auditory stimulation gait training and muscle power training (RAS-MPT) — The RAS-MPT group will attend a 60-minute training session once a week and home exercises (twice/week) for 12 weeks. Participants will receive two levels of training within each 60-minute session: (1) RAS-treadmill training and (2) MPT.
  Arms: RAS-MPT group
Behavioral: Rhythmical auditory stimulation gait training (RAS) — The RAS group will attend a 60-minute training session once a week and home exercises (twice/week) for 12 weeks. Participants will receive RAS-treadmill training repeatedly within each 60-minute session.
  Arms: RAS group
Behavioral: Muscle power training (MPT) — The MPT group will attend a 60-minute training session once a week and home exercises (twice/week) for 12 weeks. Participants will receive muscle power training repeatedly within each 60-minute session.
  Arms: MPT group
Other: Controls — Participants in the control group will receive no intervention during the study period, but continue with their normal daily activities and usual medical care. They will receive the same training as the RAS-MPT group after the study.
  Arms: Control group

SUMMARY:
Objectives: To compare the effectiveness of RAS-MPT, RAS alone, MPT alone, and usual care (as a control) for improving the overall gait performance of and reducing falls in children with developmental coordination disorder (DCD) and to explore the relationship between gait performance and falls in this population.

Design: A randomized controlled trial. Sample: 76 children with DCD. Interventions: RAS-MPT, RAS alone, MPT alone, or usual care (12 weeks). Major outcomes: Outcomes will be evaluated at baseline, post-intervention, and a 6-month follow-up. Comprehensive gait analysis will produce spatiotemporal gait parameters (e.g., velocity and stride length), kinematic gait parameters (e.g., knee joint motions), and leg muscle EMG outcomes; an isokinetic test will quantify leg muscle strength and force production time; and fall histories will be obtained via interviews. Anticipated results and significance: The RAS-MPT group is predicted to display the best gait performance, which is associated with reduced fall incidents. This novel training regime can be readily adopted in school, clinical, or home settings to improve locomotor ability in children with DCD, an outcome with positive socioeconomic implications.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 9 years old
* classified as DCD according to the Diagnostic and Statistical Manual of Mental Disorders V
* < 5th percentile on the Movement Assessment Battery for Children-2 (MABC-2)
* a total score of < 46 (for children aged 6 to 7 years 11 months) or < 55 (for children aged 8 to 9 years) on the DCD questionnaire 2007 (Chinese version)
* attending a mainstream school (i.e., intelligence level within the normal range).

Exclusion Criteria:

* any congenital, cognitive, psychiatric (e.g., comorbid attention deficit hyperactivity disorder or autism spectrum disorder), neurological, sensory, hearing, visual, vestibular, musculoskeletal, or cardiopulmonary disorder that may affect test performance
* obesity (body mass index [BMI] >95th percentile)
* receiving active treatment such as physiotherapy
* those unable to follow instructions.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in spatiotemporal gait parameter - gait velocity (m/s) | 9 months
Changes in spatiotemporal gait parameter - stride length (cm) | 9 months
Changes in spatiotemporal gait parameter - cadence (steps/min) | 9 months
Changes in spatiotemporal gait parameter - stance phase duration (% gait cycle) | 9 months
Changes in spatiotemporal gait parameter - swing phase duration (% gait cycle) | 9 months
Changes in spatiotemporal gait parameter - single-limb support durations (% gait cycle) | 9 months
Changes in spatiotemporal gait parameter - double-limb support duration (% gait cycle) | 9 months

SECONDARY OUTCOMES:
Changes in kinematic gait parameters | 9 months
  Maximum knee and ankle angles during different gait phases
Changes in leg muscle peak electromyographic values | 9 months
  Changes in leg muscle peak electromyographic values (in % of maximal voluntary isometric contraction) of rectus femoris, biceps femoris, tibialis anterior, and gastrocnemius medialis muscles
Changes in leg muscle maximum strength | 9 months
  Changes in maximum muscle strength of knee extensors and flexors and ankle plantar flexors and dorsiflexors of the dominant leg as measured by dynamometry.
Changes in leg muscle force production time | 9 months
  Changes in muscle force production time of knee extensors and flexors and ankle plantar flexors and dorsiflexors of the dominant leg as measured by dynamometry.
Changes in self-reported falls | 9 months
  Children and parents will report the number of falls within the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided